CLINICAL TRIAL: NCT03714217
Title: Weight Management in Spinal Cord Injury - Intervention and Monitoring Via Tele-Nutrition
Brief Title: Telenutrition in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-007
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injury; Obesity
Keywords: Spinal Cord Injury; Obesity; Telenutrition
MeSH Terms: conditions — Spinal Cord Injuries; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Telenutrition counseling
  Interventions: Behavioral: Telenutrition Counseling

INTERVENTIONS:
Behavioral: Telenutrition Counseling — A registered dietitian nutritionist will contact each participant twice a month for 3 months to provide nutrition counseling via iPad FaceTime.

SUMMARY:
The purpose of the study is to provide tele-nutrition counseling after a spinal cord injury (SCI). During the three months of participation, subjects will be given an iPad and the iPad will be used to record meals using a photo journal application, YouAte. In addition, subjects will receive dietary advice two times a month with a registered dietitian (RD). The dietitian role in the study will be to educate healthy weight management and accommodate any cultural and behavioral habits. The objective of this study is to show that the proposed tele-nutrition program will be effective with weight management through 3-month tele-nutrition counseling via iPad FaceTime. The hypotheses are 1) that weight and waist circumference will not increase after 3 months of tele-nutrition program, 2) quality of life will improve, and 3) quality of diet will improve.

DETAILED DESCRIPTION:
Participants with spinal cord injury (traumatic or non-traumatic) will be recruited over a 9-month period from Santa Clara Valley Medical Center's (SCVMC) inpatient rehabilitation program before discharge as well as through the outpatient SCI clinic. Demographic data, weight /height, waist circumference as well as Life Satisfaction Index-A will be obtained at enrollment and 3-months post-enrollment. For subjects unable to return to the SCVMC clinic, questionnaires will be administered over the phone and they will be asked to measure their waist circumference by themselves and with assistance from a caregiver if needed. Each participant will be provided with an iPad and 4 month cellular data plan at the time of enrollment. iPad accessories like mouthstick will be provided if needed. Prior to initiating the tele-nutrition service, each participant will be instructed on how to use the iPad and FaceTime. Registered Dietitian Nutritionist (RDN) will provide an assessment of current knowledge and nutrition evaluation at enrollment in order to individualize intervention on a per-participant basis. Counseling twice a month over a 3 month time-period via tele-nutrition using iPad FaceTime will be provided for each participant. Tele-nutrition consults, via iPad with a food photo journal application (YouAte), would emphasize the importance of tracking food intake with the primary focus on healthy weight management. Nutrition education will be tailored according to and around each individual's cultural and behavioral practice with regards to food. Participants will be counseled with the goal to make incremental changes in current diet to better optimize energy, protein, fat, and fiber intake.

YouAte, a food journaling application, will be installed on each iPad and will have a three-month membership. This app is a mindful and simple way for participants to document their food intake for the review of the RDN over the course of this project. Once a picture is taken of a meal (with assistance from a caregiver if needed), participants can choose whether they feel the meal is on-path or off-path, based on their goals. Participants can further include information about the meal in a note section if they choose to. Additional, one-tap choices of the app can further tailor each meal's mindful approach to why it was eaten, how the meal made them feel, where they ate, how it was made, and how it made them feel. RDN will be able to review all meals and snacks in order to further discuss choices and provide valuable feedback with each participant to improve intake. At the end of the 3-month participation in the tele-nutrition program, each participant will be asked to complete a satisfaction survey in addition. This app will be set up using subject identifier such as a set of numbers and/or alias. So, no Protected Health Information such as name or date of birth will be entered or used to identify the diet journaling.

Data collected throughout the study will be used to provide preliminary evidence for the feasibility of the tele-nutrition program. Baseline measures will be used to characterize the cohort and measure changes across the intervention. Quantitative changes in weight and waist circumference, as well as satisfaction survey at the end of the assessment period will be used to measure feasibility. A combination of non-parametric statistics, most likely Wilcoxon Sign Ranked Tests, and clinical assessment will be used to measure whether the changes were significant.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Traumatic or non-traumatic SCI of any level
* Is or will be living at home
* Willing to participate in a tele-nutrition program.

Exclusion Criteria:

* Medically unstable
* Unable to speak English, as the dietitian who will be providing tele-nutrition speaks only English and tele-nutrition cannot be provided with a translator
* Living in a nursing home or hospitalized at a medical facility
* Has strict dietary guidelines (e.g. diabetic, heart failure, renal, ketogenic, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline, 3 months
  Weight in kg
Change in height | Baseline, 3 months
  Height in cm
Change in waist circumference | Baseline, 3 months
  Waist circumference in cm

SECONDARY OUTCOMES:
Change in Life Satisfaction Index-A | Baseline, 3 months
  The Life Satisfaction Index A is a 20-item tool assessing quality of life. It has a total scoring range of 0 to 20, and a higher score signifies greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Shem, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No